CLINICAL TRIAL: NCT01271348
Title: Multiple-dose, Randomized, Double Blinded, Placebo-controlled, Cross Over Study of Etoricoxib for the Treatment of Muscle Pain and Inflammation Induced by Eccentric Exercise
Brief Title: Study of Etoricoxib for the Treatment of Muscle Pain and Inflammation Induced by Eccentric Exercise
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: X-pert Med GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: XPM-032
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: Muscle Pain
MeSH Terms: conditions — Myalgia | interventions — Etoricoxib

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Etoricoxib (Active Comparator)
  Interventions: Drug: Etoricoxib
- Placebo tablet (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Etoricoxib — Etoricoxib film tablet, 90 mg, q.d.
  Arms: Etoricoxib
Drug: placebo — Placebo tablet, q.d.
  Arms: Placebo tablet

SUMMARY:
Comparison of the effect of etoricoxib to placebo on muscle pain caused by eccentric contractions

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent prior to participation
* Subjects in good health as determined by the Investigator
* Age 18-40 or 50-70
* BMI > 20 and < 30
* Pain in the target muscle (thigh) during muscle contraction of at least 5 on an 11 point categorical pain rating scale
* Willing to abstain from any physical therapy, hard physical work, exercise or sauna during the study treatment periods (Screening to Final Visit)
* For females, subjects of childbearing potential (including peri-menopausal women who have had a menstrual period within 1 year) must be using appropriate birth control (defined as a method which results in a low failure rate, i.e., less than 1% per year when used consistently and correctly, such as implants, injectables, some intrauterine contraceptive devices (IUDs), sexual abstinence, or a vasectomized partner). Oral contraceptive medications are not allowed in this study. Female subjects, who are surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy) are allowed for participation

Exclusion Criteria:

* Participation in another clinical study within the last 30 days and during the study
* Subjects who are inmates of psychiatric wards, prisons, or other state institutions
* Investigator or any other team member involved directly or indirectly in the conduct of the clinical study
* Pregnancy or lactation
* Alcohol or drug abuse
* Malignancy within the past 2 years with the exception of in situ removal of basal cell carcinoma
* Known hypersensitivity to etoricoxib or other NSAID´s including Cox-2, or any of their excipients
* Bronchospasm, acute rhinitis, nasal congestion, angioneurotic edema, urticaria or allergic reactions after taking aspirin or other NSAIDs including Cox-2 inhibitors
* Major traumatic lesions (e.g. fracture, tendon or muscle ruptures) of the musculo-sceletal system of the lower limbs
* Pain conditions which might interfere with pain rating during the study, e.g. neuropathic pain
* Significant neurological or psychiatric symptoms resulting in disorientation, memory impairment, or inability to report accurately (e.g. depressive disorders, Alzheimer's disease, schizophrenia or other psychosis), that in the investigator's opinion may affect efficacy or safety assessments or may compromise subject safety during the study
* Heart failure (NYHA II-IV)
* Long term blood pressure > 140/90 mm Hg without adequate treatment
* Peripheral arterial disease, coronary heart disease and/or cerebrovascular disease
* History of stroke or myocardial infarction
* Clinically relevant ECG changes
* Estimated creatinine clearance < 60 ml/min
* Liver dysfunction (e.g. defined by ALT and/or AST levels above upper limit of normal range)
* Coagulopathy or bleeding diathesis, or concomitant use of anticoagulants including low dose aspirin
* History of pancreatitis, peptic ulcers or gastrointestinal bleedings
* Inflammatory GI disease (e.g. M. Crohn, colitis ulcerosa)
* Any other analgesic therapy including cough and cold drugs containing analgesic properties as well as any other substance used for the treatment of pain during the study observation period (Screening to final Visit)
* Any other drug that might alter pain perception like CNS active drugs
* Statins within 3 months of screening and throughout the study
* Oral anticonceptives

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pain during muscle contraction | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Rother, M.D., Study Chair — Director Clinical Operations
Locations (1):
- X-pert Med GmbH, Jena, Germany